CLINICAL TRIAL: NCT06659263
Title: A Phase 1, Open-label, Single Dose Study to Evaluate the Concentration of RE104 and Its Major Metabolites in Breast Milk and Plasma of Healthy Lactating Women.
Brief Title: RE104 Clinical Lactation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reunion Neuroscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE104-102-NHLV
Record Dates: First submitted 2024-10-14; First posted 2024-10-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-10

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 30 mg RE104 (Experimental): A single subcutaneous injection of 30 mg RE104 for Injection
  Interventions: Drug: RE104 for Injection

INTERVENTIONS:
Drug: RE104 for Injection — Single, subcutaneous dose of RE104 for Injection

SUMMARY:
The purpose of this study is to obtain data necessary to characterize the elimination of RE104 and metabolites from breastmilk of health lactating volunteers to support a regulatory assessment of when mothers can safely return to breastfeeding following a single-dose of RE104 for Injection.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 45 years of age, at least 50 kgs, and a body mass index of 18-34 kg/m2
* Has been breastfeeding or actively pumping for at least 4 weeks postpartum
* Agrees to cease breastfeeding for duration of study (Day 14) and confirms infant is able to feed from a bottle at screening.
* Willing and able to pump in order to maintain sufficient milk supply volumes for the study
* Is not pregnant or planning to become pregnant during the study
* Able to understand and adhere to study schedule and requirements and willing to sign an ICF
* In good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening

Exclusion Criteria:

* Has mastitis or other condition that would prevent the collection of milk from one or both breasts
* Active or medical history of significant mental disorder (including but not necessarily limited to major depression and anxiety disorders, bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorder and/or borderline personality disorder), or first-degree family history of psychosis or bipolar disorder
* Medically significant condition or other concomitant condition or history rendering unsuitability for the study, in the judgement of the investigator
* Has used or intends to use of prohibited medications
* Has a known sensitivity or intolerance to hallucinogenic or psychedelic substances, or potential rescue medications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to 24 hours post-dose (AUC0 24) for RE104 and 4-OH-DiPT in plasma and breast milk | Through 24 hours postdose
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for RE104 and 4-OH-DiPT in plasma and breast milk | Through 168 hours postdose
Maximum observed concentration (Cmax) for RE104 and 4-OH-DiPT in plasma and breast milk | Through 168 hours postdose
Time to reach Cmax (tmax) for RE104 and 4-OH-DiPT in plasma and breast milk | Through 168 hours postdose
Apparent total body clearance (CL/F) for RE104 in plasma | Through 168 hours postdose
Apparent volume of distribution during the terminal phase (Vz/F) for RE104 in plasma | Through 168 hours postdose
Apparent terminal elimination half-life (t1/2) for RE104 and 4-OH-DiPT in plasma | Through 168 hours postdose
Milk to plasma (M/P) ratio for RE104 and 4-OH-DiPT in breast milk | Through 168 hours postdose
Relative infant dose (RID) of RE104 and its active entity 4-OH-DiPT | Through 72 hours postdose
Total RID of RE104 and its active entity 4-OH-DiPT | Through 168 hours postdose

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) by frequency, severity and seriousness. | From dosing through study completion (post-dose follow-up is for 14 days)
  A treatment-emergent adverse event (TEAE) is defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a study drug.
Area under the concentration-time curve from time zero to 24 hours post-dose (AUC0 24) for detectable/quantifiable RE104 metabolites in plasma and breast milk | Through 24 hours postdose
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) for detectable/quantifiable RE104 metabolites in plasma and breast milk | Through 168 hours postdose
Maximum observed concentration (Cmax) for detectable/quantifiable RE104 metabolites in plasma and breast milk | Through 168 hours postdose
Time to reach Cmax (tmax) for detectable/quantifiable RE104 metabolites in plasma and breast milk | Through 168 hours postdose
Apparent terminal elimination half-life (t1/2) for detectable/quantifiable RE104 metabolites in plasma | Through 168 hours postdose
Milk to plasma (M/P) ratio for detectable/quantifiable RE104 metabolites in breast milk | Through 168 hours postdose
Amount of RE104 and its active entity 4 OH-DiPT excreted into breast milk (Ae) and amount of drug excreted into breast milk relative to dose (Fe) | Through 168 hours postdose
Unbound and bound plasma concentrations of the RE104 active entity 4-OH-DiPT. | 1, 3 and 8 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, Chief Medical Officer, Study Director — Reunion Neurosciences Inc
Locations (1):
- PPD Inc, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.